CLINICAL TRIAL: NCT00002833
Title: Use of G-CSF Stimulated HLA-Identical Allogeneic Peripheral Blood Stem Cells for Patients With High Risk Acute Myelogenous Leukemia or CML in Blast Crisis
Brief Title: Peripheral Stem Cell Transplantation Plus Filgrastim in Treating Patients With Acute or Chronic Myelogenous Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DM94-078; P30CA016672 (NIH); MDA-DM-94078 (Other: UT MD Anderson Cancer Center); NCI-G96-1001; CDR0000065035 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 1999-11-01; First posted 2004-07-30 (Estimated); Last update posted 2012-07-30 (Estimated); Status verified 2012-07

CONDITIONS: Graft Versus Host Disease; Leukemia; Myelodysplastic Syndromes
Keywords: recurrent adult acute myeloid leukemia; relapsing chronic myelogenous leukemia; chronic phase chronic myelogenous leukemia; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; adult acute myeloid leukemia in remission; Philadelphia chromosome positive chronic myelogenous leukemia; refractory anemia with excess blasts; refractory anemia with excess blasts in transformation; chronic myelomonocytic leukemia; graft versus host disease
MeSH Terms: conditions — Graft vs Host Disease; Leukemia; Myelodysplastic Syndromes; Leukemia, Myeloid, Acute; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Anemia, Refractory, with Excess of Blasts; Leukemia, Myelomonocytic, Chronic | interventions — Filgrastim; Granulocyte Colony-Stimulating Factor; Cladribine; Cyclosporine; Cytarabine; fludarabine phosphate; fludarabine; Idarubicin; Methylprednisolone; Methylprednisolone Acetate; Methylprednisolone Hemisuccinate; Peripheral Blood Stem Cell Transplantation; Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1A (Experimental): Group 1A - With or Without Remission + Failing Fludarabine therapy:
  Ara-C IV over 2 hours on days -7, -6, -5, -4 and -3 with Cladribine continuous infusion for 5 days, beginning 4 hours before Ara-C first dose. Idarubicin IV Days -6, -5 and -4. Cells infused on day 0. Cyclosporine via continuous IV infusion, oral cyclosporine administered for 6 months postinfusion (tapered 10% weekly until discontinued). Methylprednisolone begins 5 days after infusion then gradually tapered.
  Interventions: Biological: Filgrastim; Drug: Cladribine; Drug: Cyclosporine; Drug: Cytarabine (Ara-C); Drug: Idarubicin; Drug: Methylprednisolone; Procedure: Peripheral Blood Stem Cell Transplantation
- Group 1B (Experimental): Group 1B: With or Without Remission, No previous Fludara Therapy
  Fludarabine IV over 30 minutes daily on days -6, -5, -4 and -3. Ara-C IV begins 4 hours after fludarabine infusion, continues for 4 hours. Idarubicin IV Days -6, -5 and -4. Cells infused on day 0. Cyclosporine via continuous IV infusion, oral cyclosporine administered for 6 months postinfusion (tapered 10% weekly until discontinued). Methylprednisolone begins 5 days after infusion then gradually tapered.
  Interventions: Biological: Filgrastim; Drug: Cyclosporine; Drug: Cytarabine (Ara-C); Drug: Fludarabine Phosphate; Drug: Idarubicin; Drug: Methylprednisolone; Procedure: Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Biological: Filgrastim — Donors receive Filgrastim SC (Subcutaneously) every 12 hours for 2 days prior to stem cell collection.
  Other Names: G-CSF; Neupogen
Drug: Cladribine — Continuous infusion for 5 days, beginning 4 hours before Ara-C first dose.
  Other Names: Leustatin; 2-CdA
  Arms: Group 1A
Drug: Cyclosporine — For GVHD prophylaxis, cyclosporine via continuous IV infusion. Oral cyclosporine administered once tolerating oral feeding and continued for 6 months postinfusion. Then dose tapered 10% weekly until discontinued.
  Other Names: Sandimmune; CYA; Cyclosporin A
Drug: Cytarabine (Ara-C) — Group 1A: Ara-C IV over 2 hours on days -7, -6, -5, -4 and -3; Group 1B: Ara-C IV begins 4 hours after fludarabine infusion, continues for 4 hours.
  Other Names: Ara-C; Cytosar; DepoCyt; Cytosine Arabinosine Hydrochloride
Drug: Fludarabine Phosphate — IV over 30 minutes daily on days -6, -5, -4 and -3.
  Other Names: Fludara; Fludarabine
  Arms: Group 1B
Drug: Idarubicin — IV Days -6, -5 and -4.
  Other Names: Idamycin
Drug: Methylprednisolone — Begins 5 days after infusion and is gradually tapered.
  Other Names: Depo-Medrol; Medrol; Solu-Medrol
Procedure: Peripheral Blood Stem Cell Transplantation — Cell infusion Day 0.
  Other Names: PBSCT; Stem Cell Transplant

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining chemotherapy with peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more cancer cells. Colony stimulating factors such as filgrastim may increase the number of immune cells found in bone marrow or peripheral blood and may help a person's immune system recover from the side effects of chemotherapy.

PURPOSE: Phase II trial to study the effectiveness of peripheral stem cell transplantation plus filgrastim in treating patients who have acute or chronic myelogenous leukemia.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the toxic effects and feasibility of using filgrastim in promoting hematopoietic recovery and leukemia control after intensive but nonmyeloablative salvage chemotherapy. II. Determine the engraftment kinetics and degree of chimerism achievable.

OUTLINE: The trial will have 2 patient groups. Patients not in remission are assigned to group 1, while patients in remission are assigned to group 2. Then, groups are divided into 2 treatment arms. Patients failing fludarabine therapy receive cytarabine (Ara-C) IV over 2 hours on days -7, -6, -5, -4 and -3. Beginning 4 hours before the first dose of Ara-C, patients receive cladribine (2-chlorodeoxyadenosine; 2-CdA) by continuous infusion for 5 days. Patients without prior fludarabine therapy receive fludarabine IV over 30 minutes daily on days -6, -5, -4 and -3. Ara-C IV begins 4 hours after the beginning of the fludarabine infusion and continues for 4 hours. Idarubicin IV is given on days -6, -5 and -4. Donors receive filgrastim SC every 12 hours for 2 days prior to stem cell collection. Cells are infused on day 0. For GVHD prophylaxis, all patients receive cyclosporine via continuous IV infusion. Oral cyclosporine is administered once patients tolerate oral feeding and continued for 6 months postinfusion. Then, the dose of cyclosporine is tapered 10% weekly until discontinued. Methylprednisolone begins 5 days after infusion and is gradually tapered.

PROJECTED ACCRUAL: A maximum of 15 patients per arm are likely to be entered in 24 to 36 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Acute leukemia with poor risk cytogenetic features (-5,-7, +8) in first complete remission Poor risk myelodysplasia Refractory anemia with excess blasts (RAEB) RAEB in transformation (RAEB-T) Chronic myelomonocytic leukemia (CMML) Chronic myelogenous leukemia (CML) in late chronic phase Acute leukemia with greater than first complete remission or transformed CML or CMML

PATIENT CHARACTERISTICS: Age: 55 to 65 65 to 70 (at the discretion of study chairperson on basis of performance status) 55 and under (if declined for conventional high dose chemotherapy due to concurrent medical conditions (i.e. ejection fraction less than 50, FEV1, FVC, or DLCO less than 50%, abnormal LFTs) Performance status: Zubrod less than 2 Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Bilirubin less than 3 mg/dL Renal: Serum creatinine less than 2 mg/dL Cardiovascular: Ejection fraction greater than 40% per MUGA scan Pulmonary: Not specified Other: No active uncontrolled infection HLA compatible donor capable of donating stem cells via apheresis

PRIOR CONCURRENT THERAPY: Not specified

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 1994-10; Primary Completion 2002-04 (Actual); Study Completion 2002-04 (Actual)

PRIMARY OUTCOMES:
Toxic Effects of Peripheral Stem Cell Transplantation + Filgrastim | 24 - 36 months
  Effectiveness as determined by toxic effects and feasibility of using filgrastim in promoting hematopoietic recovery and leukemia control after intensive but nonmyeloablative salvage chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Giralt, MD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas - MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center — http://www.mdanderson.org